CLINICAL TRIAL: NCT02590588
Title: Study of Phosphatidylinositol-3-kinase (PI3K) Inhibitor, Idelalisib (GS-1101), in IgM-Associated AL Amyloid
Brief Title: Idelalisib for Immunoglobulin M (IgM)-Associated Primary (AL) Amyloidosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: John Mark Sloan (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, John Mark Sloan, Associate Professor of Medicine, Boston Medical Center
Organization: Boston Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-34318
Record Dates: First submitted 2015-09-09; First posted 2015-10-29 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Amyloidosis
Keywords: IgM-associated AL amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idelalisib (Experimental): Idelalisib 100 mg twice daily with possible escalation after 3 months to 150 mg twice daily at investigator discretion.
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib daily until unacceptable toxicity or disease progression.
  Other Names: GS-1101

SUMMARY:
The investigators expect to enroll 15 participants with relapsed or refractory IgM-associated AL amyloidosis onto this Phase II clinical trial. Idelalisib will be self-administered orally at a dose of 100 mg twice daily (may be increased to 150 mg (one tablet) twice daily after 3 months at investigator discretion). Participants will be treated until disease progression, unacceptable toxicity, or decision to withdraw from the trial. Disease evaluations will be performed every three months until disease progression.

DETAILED DESCRIPTION:
This study includes the use of Idelalisib to treat previously treated patients with IgM-associated AL Amyloidosis at Boston Medical Center. Boston Medical Center is internationally recognized as a leader in amyloidosis research and patient care through the activities of the multidisciplinary Amyloid Center at Boston University. The problematic cell in most forms of AL amyloidosis shares similarities with multiple myeloma. However, in the small subset of AL Amyloidosis patients with an IgM paraprotein, the cells are more typically related to lymphoplasmacytic lymphoma or Waldenstrom's macroglobulinemia. Because clonal cluster of differentiation antigen 20 (CD20)+ lymphoplasmacytic cells are usually responsible for IgM paraproteins, treatment paradigms based on Waldenstrom's macroglobulinemia (WM) may be more appropriate than myeloma-based strategies. Idelalisib has been shown to be active and well tolerated in patients with relapsed/refractory non-Hodgkin lymphoma including chronic lymphocytic lymphoma, and lymphoplasmacytic lymphoma with or without Waldenström's macroglobulinemia (WM). The side effect profile of idelalisib merges well with the known predisposition to toxicity of amyloidosis patient.

The investigators expect to enroll 15 participants with IgM-associated AL amyloidosis onto this Phase II clinical trial. Idelalisib will be self-administered orally at a dose of 100 mg (1 tablet) twice daily (may be escalated to 150 mg (one tablet) twice daily after 3 months at investigator discretion). Participants will be treated until disease progression, unacceptable toxicity, or decision to withdraw from the trial. Disease evaluations will be performed every three months until disease progression.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 IgM paraprotein identified on serum immunofixation electrophoresis OR light chain-restricted CD20+ lymphoplasmacytic population on biopsy of bone marrow or lymph node (identified by H&E/immunohistochemistry or flow cytometry) OR positive myeloid differentiation primary response gene 88 (MYD88-L265P) OR CXCR4WHIM mutation (CXCR4 mutation - warts, hypogammaglobulinemia, infections, myelokathexis) on submitted samples

3.1.2 Biopsy-proven relapsed or refractory AL amyloidosis

3.1.3 Age ≥ 18 years

3.1.4 Eastern Cooperative Oncology Group (ECOG) performance status <2 (see Appendix A.)

3.1.5 Difference between serum free light chains (FLC) of >30 mg/L or quantifiable IgM paraprotein >0.5 g/L

3.1.6 Participants must have normal organ and marrow function as defined below:

* Absolute neutrophil count > 1,000/mm3
* Platelets > 50,000/mm3

3.1.7 Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

3.2.1 Previous treatment with idelalisib

3.2.2 Glomerular filtration rate (GFR) <15 ml/min

3.2.3 Cardiac biomarker Stage III disease as determined by B-type natriuretic peptide (BNP) >100 pg/mL and Troponin-I >0.1 ng/mL (Girnius 2014)

3.2.4 alanine-aminotransferase (ALT)/aspartate aminotransferase (AST) values >2.5x upper limit of normal, Bilirubin >1.5 upper limit of normal (ULN)

3.2.5 Central nervous system (CNS) malignancy or other active malignancy

3.2.6 Lactating or pregnant women

3.2.7 Exposure to another investigational drug within 4 weeks prior to start of study treatment

3.2.8 Ongoing alcohol or drug addiction as determined by investigator

3.2.9 Amyloid-directed therapy within the past 28 days

3.2.10 History of Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV) (assessed by positive Hepatitis B polymerase chain reaction assay (PCR) or Hepatitis B Surface Antigen), and/or Hepatitis C Virus (HCV) infection

3.2.11 t(11,14) translocation identified on bone marrow cytogenetics or by Fluorescence in situ hybridization (FISH)

3.2.12 Known lytic bone lesions

3.2.13 Positive cytomegaly virus (CMV) Polymerase chain reaction (PCR)

3.2.14 Previously untreated AL amyloidosis (Newly diagnosed)

3.2.15 Unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John "Mark" Sloan, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Idelalisib
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 'There was only one patient enrolled
Units Other Than Participants: only patient enrolled
Arm/Group | Idelalisib
Number analyzed (Participants) | 1
Number analyzed (only patient enrolled) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Unit of measure based on patient identification
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 1
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Evaluate hematologic response according to standard criteria
Time Frame: 3 months
Population: Number of participants with hematologic response is zero. There was only one patient enrolled and he did not remain on study long enough for his first 3 month response evaluation.
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival
Description: Evaluate time to progression
Time Frame: 1 year
Population: The evaluation of progression-free survival requires that a patient responds, and then progresses. There was only one patient enrolled and he did not remain on study long enough for his first 3 month response evaluation.
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

3. Secondary Outcome: Organ Response
Description: Number of patients with organ response using standard AL amyloidosis criteria.
Time Frame: 3 months
Population: Number of patients with organ response using standard AL amyloidosis criteria.
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

4. Secondary Outcome: Evaluate Safety and Tolerability of Agent
Description: Number of Participants With Treatment-Related Adverse Events as Assessed by Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0
Time Frame: 3 months
Population: There was only one patient enrolled and he did experience treatment-related adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Quality of Life
Description: Evaluate quality of life according to Functional Assessment of Cancer Therapy Lymphoma Subscale (FACT-Lym) assessment tool
Time Frame: 3 months
Population: 'There was only one patient enrolled and he did not remain on study long enough for his first protocol-specified quality of life assessment
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Idelalisib
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idelalisib (N=1)
increased (Investigations) | 1 (1) — alanine-aminotransferase
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idelalisib (N=1)
nausea (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
diminished appetite (Gastrointestinal disorders) | 1 (1)
swollen eyelids (Eye disorders) | 1 (1)
discolored urine (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT02590588/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT02590588/ICF_001.pdf